CLINICAL TRIAL: NCT03187626
Title: Short-term Efficacy of a Single Ultrasound-guided Intra-articular Injection of Botulinum Toxin A Associated With Splinting for Base-of-thumb Osteoarthritis: a Randomized Controlled Double-blind Pilot Study
Brief Title: Efficacy of an Intra-articular Injection of Botulinum Toxin A Associated With Splinting for Base-of-thumb Osteoarthritis
Acronym: RHIBOT
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P160404
Record Dates: First submitted 2017-06-13; First posted 2017-06-15 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Base-of-thumb Osteoarthritis
Keywords: Base-of-thumb osteoarthritis; Botulinum toxin A; Intra-articular therapy; Randomized trial
MeSH Terms: interventions — Botulinum Toxins, Type A; Idoxuridine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intra-articular botulinum toxin A and splinting (Experimental): Ultrasound-guided injection of 50 Allergan Unities of botulinum toxin A (Botox®, Allergan) resuspended in 1 ml of saline in the trapeziometacarpal joint and custom-made thermoformed plastic splint to be worn for 48 hours after intra-articular injection then nightly
  Interventions: Drug: botulinum toxin A
- Intra-articular saline and splinting (Active Comparator): Ultrasound-guided injection of 1 ml of saline in the trapeziometacarpal joint and custom-made thermoformed plastic splint to be worn for 48 hours after intra-articular injection then nightly
  Interventions: Drug: saline

INTERVENTIONS:
Drug: botulinum toxin A — Ultrasound-guided injection of 50 Allergan Unities of botulinum toxin A (Botox®, Allergan) resuspended in 1 ml of saline in the trapeziometacarpal joint and custom-made thermoformed plastic splint to be worn for 48 hours after intra-articular injection then nightly
  Other Names: Botox®; Allergan
  Arms: Intra-articular botulinum toxin A and splinting
Drug: saline — Ultrasound-guided injection of 1 ml of saline in the trapeziometacarpal joint and custom-made thermoformed plastic splint to be worn for 48 hours after intra-articular injection then nightly
  Arms: Intra-articular saline and splinting

SUMMARY:
The primary purpose of this study is to determine whether a single ultrasound-guided intra-articular injection of botulinum toxin A associated to splinting is effective in reducing pain at 3 months in base-of-thumb osteoarthritis.

DETAILED DESCRIPTION:
Base-of-thumb osteoarthritis is a common condition affecting middle-age persons. Base-of-thumb osteoarthritis induces pain and hand-specific limitations in activities. For short and midterm effects, therapeutic options usually include splinting, exercise therapy and intra-articular injections of glucocorticoids or hyaluronic acid. However, evidence of efficacy of intra-articular therapies in base-of-thumb osteoarthritis and international guidelines are inconsistent. Recently, the use of intra-articular botulinum toxin A as a pain killer has raised intense interest. The exact mechanisms of pain modulation by botulinum toxin A in osteoarthritis are unclear. It has been suggested that botulinum toxin A could directly reduce peripheral sensitization and indirectly reduce central sensitization. Indeed, recent studies suggest an inhibitory role of botulinum toxin A on the release of mediators involved in nociception, such as P substance, calcitonin gene-related peptide and glutamate. Open and randomized controlled trials of botulinum toxin A in knee osteoarthritis support short to mid-term positive clinical effects on pain. However, no study has reported results for base-of-thumb osteoarthritis

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Pain intensity on a self-administered 11-point pain numeric rating scale ≥ 30
* Pain involving the base-of-thumb
* X-ray evidence of base-of-thumb osteoarthritis with at least 2 of the 4 following items involving the trapeziometacarpal joint : osteophytes, joint space narrowing, subchondral bone sclerosis or subchondral cysts
* 1990 American College of Rheumatology classification criteria for hand osteoarthritis adapted to base-of-thumb osteoarthritis
* Medical examination
* Written consent
* Health insurance
* For women of childbearing age, a negative urinary pregnancy test

Exclusion Criteria:

* History of thumb surgery
* History of inflammatory or crystal-associated rheumatic disease
* Neurological disorders involving the hands other than carpien canal syndrom
* Collagen disorders involving the hands : Dupuytren, Marfan or Ehlers-Danlos diseases
* Osteoarthritis predominating at the scaphotrapezial joint on X-Ray
* Hand or wrist trauma ≤ 2 months
* Hand or wrist intra-articular injections ≤ 2 months
* Contra-indication to botulinum toxin A injection or to splinting
* Cognitive or behavioral disorders making the assessment impossible
* Participant unable to speak, read and write french
* Bilateral BTOA without predominant symptomatic side
* Pregnancy and breast feeding
* Persons referred to in Articles L 1121-5; 6; 8; 9 of the Public Health Code (protected minors or adults, guardianship or trusteeship, etc.)
* Patient with epilepsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-11-29 (Actual); Primary Completion 2021-02-16 (Actual); Study Completion 2021-04-23 (Actual)

PRIMARY OUTCOMES:
Change in base-of-thumb pain 3 months post-injection | 3 months post injection
  Mean change from baseline in average base-of-thumb pain intensity in the previous 48 hrs on a self-administered 11-point pain numeric rating scale (0 no pain - 100 maximal pain)

SECONDARY OUTCOMES:
Change in base-of-thumb pain 1 month post-injection | 1 month post injection
  Mean change from baseline in average base-of-thumb pain intensity in the previous 48 hrs on a self-administered 11-point pain numeric rating scale (0 no pain - 100 maximal pain)
Change in base-of-thumb pain 6 months post-injection | 6 months post injection
  Mean change from baseline in average base-of-thumb pain intensity in the previous 48 hrs on a self-administered 11-point pain numeric rating scale (0 no pain - 100 maximal pain)
Change in hand function 3 months post-injection | 3 months post injection
  Mean change from baseline in average hand-specific limitations in activities in the previous 2 weeks on the self-administered Cochin Hand Function Scale (0 no limitations - 90 maximal limitations)
Change in hand function 6 months post-injection | 6 months post injection
  Mean change from baseline in average hand-specific limitations in activities in the previous 2 weeks on the self-administered Cochin Hand Function Scale (0 no limitations - 90 maximal limitations)
Change in patient's global assessment 3 months post-injection | 3 months post-injection
  Mean change from baseline in patient's global assessment on a self-administered 11-point numeric rating scale (0 worst possible - 100 best possible)
Change in patient's global assessment 6 months post-injection | 6 months post-injection
  Mean change from baseline in patient's global assessment on a self-administered 11-point numeric rating scale (0 worst possible - 100 best possible)
Percentage of OARSI responders 3 months post-injection | 3 months post-injection
  OARSI response is defined as an improvement in pain (0 to 100 numeric rating scale) or in function (0 to 90 Cochin Hand Function Scale) ≥ 50% and absolute change ≥ 20/100 on pain numeric rating scale or ≥ 9/90 on Cochin Hand Function Scale respectively , or improvement in at least 2 of the 3 following items: 1/ pain ≥ 20% and absolute change ≥ 10/100, 2/ function ≥ 20% and absolute change ≥ 9/90, 3/ patient's global assessment (0 to 100 numeric rating scale) ≥ 20% and absolute change ≥ 10/100
Percentage of OARSI responders 6 months post-injection | 6 months post-injection
  OARSI response is defined as an improvement in pain (0 to 100 numeric rating scale) or in function (0 to 90 Cochin Hand Function Scale) ≥ 50% and absolute change ≥ 20/100 on pain numeric rating scale or ≥ 9/90 on Cochin Hand Function Scale respectively , or improvement in at least 2 of the 3 following items: 1/ pain ≥ 20% and absolute change ≥ 10/100, 2/ function ≥ 20% and absolute change ≥ 9/90, 3/ patient's global assessment (0 to 100 numeric rating scale) ≥ 20% and absolute change ≥ 10/100
Analgesics consumption at 3 months | from injection to 3 months post-injection
  Self-reported consumption of analgesics (non-opioid, weak and strong opioids) using a self-administered 4-class scale (never; several times a month; several times a week; daily)
Analgesics consumption at 6 months | from 3 to 6 months post-injection
  Self-reported consumption of analgesics (non-opioid, weak and strong opioids) using a self-administered 4-class scale (never; several times a month; several times a week; daily)
Non-steroidal anti-inflammatory drugs consumption at 3 months | from injection to 3 months post-injection
  Self-reported consumption of non-steroidal anti-inflammatory drugs using a self-administered 4-class scale (never; several times a month; several times a week; daily)
Non-steroidal anti-inflammatory drugs consumption at 6 months | from 3 to 6 months post-injection
  Self-reported consumption of non-steroidal anti-inflammatory drugs using a self-administered 4-class scale (never; several times a month; several times a week; daily)

CONTACTS AND LOCATIONS:
Overall Officials: François RANNOU, MD, PhD, Study Director — AP-HP , université Paris Descartes; Christelle NGUYEN, MD, PhD, Principal Investigator — AP-HP, université Paris Descartes
Locations (1):
- Assistance Publique - Hôpitaux de Paris, Service de Rééducation et de Réadaptation de l'Appareil Locomoteur et des Pathologies du Rachis, Hôpital Cochin, Paris, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gil C, Abdoul H, Campagna R, Guerini H, Ieong E, Chagny F, Bedin C, Roren A, Lefevre-Colau MM, Poiraudeau S, Feydy A, Rannou F, Nguyen C. Intra-articular botulinum toxin A for base-of-thumb osteoarthritis: protocol for a randomised trial (RHIBOT). BMJ Open. 2018 Jun 30;8(6):e022337. doi: 10.1136/bmjopen-2018-022337. PMID 29961037
- [Derived] Nguyen C, Abdoul H, Campagna R, Guerini H, Jilet L, Bedin C, Chagny F, Couraud G, Daste C, Drape JL, Flechon R, Gil C, Guerin C, Lefevre-Colau MM, Poiraudeau S, Randriamampandry E, Roren A, Feydy A, Rannou F. Intra-articular botulinum toxin A injection for painful base-of-thumb osteoarthritis: a double-blind, randomised, controlled, phase 3 trial (RHIBOT). Lancet Rheumatol. 2022 Jul;4(7):e480-e489. doi: 10.1016/S2665-9913(22)00129-1. PMID 38294016